CLINICAL TRIAL: NCT03497663
Title: VIA Family - Family Based Early Intervention Versus Treatment as Usual. Study Protocol for a Randomized Clinical Trial. Can a Multidisciplinary Specialized Intervention Improve General Functioning and Decrease Symptoms of Psychopathology in Familial High Risk Children Born to Parents With Severe Mental Illness?
Brief Title: VIA Family - Family Based Early Intervention Versus Treatment as Usual
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Municipality of Frederiksberg, Denmark (Unknown); Ministry of the Interior and Health, Denmark (Other Government); TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIAFAMILYFEB18
Record Dates: First submitted 2018-03-19; First posted 2018-04-13 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2020-10

CONDITIONS: Early Intervention; Child of Impaired Parents; Child; Adolescent; Mental Disorders, Severe; Schizophrenia; Bipolar Disorder; Depressive Disorder, Recurrent; Psychotic Disorders; Parent-Child Relations
Keywords: Familial high risk; offspring; schizophrenia; bipolar disorder; recurrent depression; early intervention; parental training; family based intervention
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Depressive Disorder; Recurrence; Psychotic Disorders; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The families randomly assigned to the VIA Family Group will be offered regular contact with a case manager. A multidisciplinary team of specialists from adult mental health services/psychiatry , child and adolescent mental health services and social services will be responsible for providing the basic treatment elements that are: case management, psychoeducation for the whole family, parental training (Triple P) and early intervention for mental problems of the child.
Who Masked: Outcomes Assessor
Masking Description: Baseline Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIA Family intervention (Experimental): VIA Family is a family based intervention. A multidisciplinary team of specialists from adult mental health services, child and adolescent mental health services and social services will be responsible for providing the basic treatment elements that are: case management and regular contact with the case manager, psychoeducation for the whole family, parental training (Triple P) and early intervention for mental problems of the child.
  Interventions: Other: VIA Family intervention
- Treatment as Usual (TAU) (Active Comparator): TAU is defined as any kind of help and support focusing on high risk children and parental mental illness. At present, the municipalities and the mental health services do not offer any kind of family focused intervention addressing parental mental illness that can be compared to the VIA Family program.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Other: VIA Family intervention — Family based intervention
  Arms: VIA Family intervention
Other: Treatment As Usual — Treatment As Usual
  Other Names: TAU
  Arms: Treatment as Usual (TAU)

SUMMARY:
This RCT aims to investigate the effect of an early family-based intervention (VIA Family) focusing on reducing risk and increasing resilience for children in families where at least one parent has a severe mental illness.The study is a randomized clinical trial including 100 children age 6-12 with familial high risk.The children and their parents will be assessed at baseline and thereafter randomized and allocated to either Treatment as Usual or VIA Family.

DETAILED DESCRIPTION:
Background: Children born to parents with severe mental illness like schizophrenia, bipolar disorder or major recurrent depression have an increased risk of developing a mental illness themselves during life. These children are also more likely to display developmental delays, cognitive disabilities, social problems and may have a higher risk than background population of experiencing adverse life events. This is due to both genetic and environmental factors, but in spite of the well documented increased risk for children with familial high risk no family-based early intervention has been developed. This study aims to investigate the effect of an early intervention model focusing on reducing risk and increasing resilience for children in families where at least one parent has a severe mental illness.

Methods: The study is a randomized clinical trial including 100 children age 6-12 with familial high risk. Families will be recruited from registers or be referred from the primary sector or from hospitals. The children and their parents will be assessed at baseline and thereafter randomized and allocated to either Treatment as Usual or VIA Family. In the VIA Family group the families will be offered regular contact with a case manager. A multidisciplinary team of specialists from Adult Mental Health Services, Child and Adolescent Mental Health Services and Social Services will be responsible for providing the basic treatment elements that are: case management, psychoeducation for the whole family, parental training (Triple P) and early intervention for mental problems of the child. The study period is 18 months for both groups and all participants will be assessed at baseline and after 18 months. Primary outcome measure will be daily functioning of the child (CGAS), and secondary measures are psychopathology in the child and days of school absence, family functioning and child's home environment.

Discussion: This study is to the investigators knowledge the first to explore the effects on children with familial high risk for severe mental illness of a multidisciplinary team intervention providing an intensive and flexible support matching the families' needs. The study will provide important knowledge about the possibilities of increasing resilience and reducing risk of a child by supporting the whole family. However, longer follow-up time may be needed.

ELIGIBILITY:
Inclusion Criteria:

* Child must have address registered in the municipality of Frederiksberg or Copenhagen.
* At least one of the biological parents must have a diagnosis of schizophrenia spectrum disorder, bipolar affective disorder or recurrent major depression.
* The parent with a diagnosis must have had at least one in- or outpatient contact with the mental health system within the lifetime of the child.

Exclusion Criteria:

* Parents who do not speak and understand enough Danish to be able to give informed consent for their own and for the child's participation.
* If all family members are currently engaged in an intensive family intervention program addressing parental functioning and child development, they are excluded from the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Childrens Global Assesment Scale (CGAS) | Change from baseline at 18 month follow-up
  A clinician rated measurment to asses general functioning in children (scale from 1-100. High score represent better outcome)

SECONDARY OUTCOMES:
Change in Childrens Behaviour Checklist (CBCL) | Change from baseline at 18 month follow-up
  Parent and teacher reported questionaire on child behavior ( low score represent better outcome).
Change in Family Assessment Device (FAD) | Change from baseline at 18 month follow-up
  A 60 item parent report questionaire assesing family functioning ( scale 1-4. Low score represent better outcome)
Change in child's number of days absent from school | Change from baseline at 18 month follow-up
  Number of days child was absent from school within the last 6 month (low number represent better outcome). Teacher rated.
Change in Home Observation for Measurement of the Environment (HOME) | Change from baseline at 18 month follow-up
  A clinican rated semi structured interview measuring stimulation and support in the home ( scale 0-60. High score represent better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Thorup, Principal Investigator — Research Unit at Child and Adolescent Mental Health Center, Capital Region, Denmark
Locations (1):
- Research Unit at Child and Adolescent Mental Health Center, Capital Region, Copenhagen, Denmark

REFERENCES:
- [Derived] Muller AD, Gjode ICT, Christensen SH, Jorgensen SK, Fischer K, Moszkowicz M, Hemager N, Nordentoft M, Piche G, Thorup AAE. Perceived Need and Social Relatedness Contribute to Change in Selective Prevention for Mental Illness: a Mixed Methods Study. Prev Sci. 2025 Aug;26(6):908-920. doi: 10.1007/s11121-025-01831-w. Epub 2025 Aug 12. PMID 40796986
- [Derived] Gjode ICT, Muller AD, Hjorthoj C, Hemager N, Ingversen S, Moszkowicz M, Christensen SH, Mikkelsen LJ, Nielsen SS, Melau M, Forman J, Nordentoft M, Thorup AAE. Effects on family functioning and the home environment of a family-based preventive intervention for children of parents with severe mental illness: A randomized controlled trial. J Consult Clin Psychol. 2025 Apr;93(4):267-280. doi: 10.1037/ccp0000924. Epub 2024 Dec 12. PMID 39666517
- [Derived] Muller AD, Gjode ICT, Eigil MS, Busck H, Bonne M, Nordentoft M, Thorup AAE. VIA Family-a family-based early intervention versus treatment as usual for familial high-risk children: a study protocol for a randomized clinical trial. Trials. 2019 Feb 8;20(1):112. doi: 10.1186/s13063-019-3191-0. PMID 30736834

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT03497663/SAP_000.pdf